CLINICAL TRIAL: NCT04699695
Title: A Prospective Multicenter Sample Collection Study Using Non-invasive Methods to Investigate Biomarkers in Pediatric and Adult Patients With Atopic Dermatitis
Brief Title: A Prospective Sample Collection Study Using Non-invasive Methods to Investigate Biomarkers in AD Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: DermTech (Other)
Responsible Party: Sponsor
Other Study IDs: DermTech 20-03
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-03

CONDITIONS: Atopic Dermatitis
Keywords: DermTech; Biologics
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — samples collected non-invasively will be assess for nucleic acids and microbiome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Biologic Treatment: Subjects prescribed a biologic agent per standard of care
  Interventions: Other: Biologic therapy versus no biologic therapy
- Other Treatments: Subjects prescribed other treatment modalities exclusive of biologic therapy per standard of care
  Interventions: Other: Biologic therapy versus no biologic therapy

INTERVENTIONS:
Other: Biologic therapy versus no biologic therapy — Biologic therapy administered per standard of care

SUMMARY:
This is a prospective, multicenter, sample collection study using DermTech's non-invasive skin collection kits to evaluate genomic biomarkers and microbiome information from pediatric and adult subjects with atopic dermatitis(AD). Samples collected will be analyzed to detect gene signatures and microbiome populations associated with AD and sub-populations of AD.

DETAILED DESCRIPTION:
This is a prospective, multicenter, sample collection study using DermTech's non-invasive skin collection kits to evaluate genomic biomarkers and microbiome information from pediatric and adult subjects with atopic dermatitis. Samples collected will be analyzed to detect gene signatures and microbiome populations associated with atopic dermatitis and sub-populations of AD.

Approximately 500 pediatric and adult subjects with moderate to severe AD will be enrolled in this study. Non-invasive skin samples will be collected at baseline, before drug administration 16 weeks (+/- 2 weeks) after treatment with biological therapy and a final visit at 26 weeks ((+/- 4 weeks).

Subjects will enter the Screening Period once the informed consent and/or assent process has been completed.

Once patient eligibility is confirmed, non-invasive skin samples will be collected using DermTech's non-invasive sample collection kit.

Samples will be collected from the following areas:

* Target Lesion - lesional skin for genomic analysis. Please note the location for subsequent collections.
* Lesional skin for microbiome analysis similar in size and severity to the target lesion noted above. Please note the location for subsequent collections.
* Non-lesional skin at least 5 cm from any active lesion. The intervals for subsequent sample collection, if applicable, will be determined based on standard of care (SOC) treatment and the subject's willingness to undergo repeat non-invasive sampling.

Data to be collected includes eczema area and severity index (EASI), patient oriented eczema measure (POEM), investigator global assessment (IGA), peak pruritus numerical rating scale (PPNRS), and transepidermal water loss (TEWL).

Photographic documentation of the site(s) sampled should be obtained to confirm consistent sampling of the lesional and non-lesional sites. Each non-invasive sample collection will consist of sequential application of 4 individual patches to a site. If during active treatment the skin lesion disappears during active treatment, skin samples will still be obtained from the same location.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females at least 1 year of age;
2. Subjects with documented, active moderate to severe atopic dermatitis;
3. Subjects must have a history of atopic dermatitis for at least three months;
4. Subjects with no known reactions to adhesives;
5. Subject has a sufficient number of target plaques on the central body, which includes knees or elbows, and not limited to lesions on the mucosal membranes, soles of the feet or palms of the hands;
6. Subjects willing to follow standard of care (SOC) for his/her atopic dermatitis; and
7. Subjects must be able to complete all study visits required by the protocol.

Exclusion Criteria:

1. Pregnant or breast feeding, including positive pregnancy test at baseline or expected to become pregnant during participation in the trial;
2. History of cancer (exceptions for: a) non-metastatic malignancy deemed cured at the time of enrollment, b) skin cancer that has been excised with controlled margins or has not recurred in 6 months; and c) treated cervical cancer in situ);
3. Current acute infectious illness (viral, parasitic or bacterial) within 4 weeks of enrollment;
4. Receipt of systemic anti-atopic dermatitis medication, including retinoids, corticosteroids, cyclosporine, methotrexate within the four weeks of the Baseline Visit;
5. Use of topical therapy (except emollients) for atopic dermatitis or any other condition within two weeks of the Baseline Visit;
6. Receipt of any investigational drug therapy within four weeks or 5 half-lives, whichever is longer of study enrollment, or concurrent participation in another interventional clinical study; and
7. Documented substance abuse, any other significant medical condition or laboratory result that would indicate an unreasonable risk to the subject or potential interference with study procedures, or would negatively affect the patient's reliability and compliance with the study schedule.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 500 pediatric and adult subjects with moderate to severe atopic dermatitis will be enrolled in this study
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Gene expression with primary disease assessment EASI | Week 16
  Expression of genes with disease activity measures including the EASI score

SECONDARY OUTCOMES:
Gene expression correlated with POEM assessment | Week 16
  Expression of genes in the DermTech assay with POEM disease activity
Gene expression correlated with IGA assessment | Week 16
  Expression of genes in the DermTech assay with IGA disease activity
Gene expression correlated with TEWL assessment | Week 16
  Expression of genes in the DermTech assay with TEWL
Gene expression correlated with PRNS assessment | Week 16
  Expression of genes in the DermTech asssay with PPRNS

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Orit Markowitz, New York, New York
  - Lisa A. Beck, Rochester, New York

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared with other researchers and patient data will be de-identified.

REFERENCES:
- [Background] Yao Z, Moy R, Allen T, Jansen B. An Adhesive Patch-Based Skin Biopsy Device for Molecular Diagnostics and Skin Microbiome Studies. J Drugs Dermatol. 2017 Oct 1;16(10):979-986. PMID 29036251